CLINICAL TRIAL: NCT06432790
Title: Comparative-effectiveness of a Healthy Lifestyle and Asthma Management Program, In-person vs. ONline (CHAMPION)
Brief Title: Comparative-effectiveness of a Healthy Lifestyle and Asthma Management Program, In-person vs. ONline
Acronym: CHAMPION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Lauren G. Fiechtner, M.D., Assistant Professor of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2024P001418; TE-2022C3-30362 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Overweight, Childhood; Obesity, Childhood; Asthma in Children
Keywords: telehealth
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHAMPION via Telehealth (Experimental): * Intensive 0-6 months: 1 individual visit monthly (virtual), 1 group visit monthly (virtual)
  * Maintenance 6-12 months: 1 individual visit monthly (virtual), 2 health coaching calls per month
  Interventions: Behavioral: CHAMPION
- CHAMPION via In-Person (Active Comparator): * Intensive 0-6 months: 1 individual visit monthly (in-person), 1 group visit monthly (in-person)
  * Maintenance 6-12 months: 1 individual visit monthly (in-person), 2 health coaching calls per month
  Interventions: Behavioral: CHAMPION

INTERVENTIONS:
Behavioral: CHAMPION — The CHAMPION program is an intensive health behavior and lifestyle treatment (IHBLT), formed through the integration of the Healthy Weight Clinic IHBLT and with MGB's pediatric Asthma Population Health Management Program. It consists of 30 hours of contact time with the CHAMPION team (physician, dietician, community health worker), consistent with the USPSTF and AAP recommendations, monthly individual clinic visits with the team (in person or virtual, per randomization), health coaching calls with a community health worker and/or registered dietician, monthly group sessions (in the first six months), and educational materials for families that reinforce healthy lifestyle behaviors and provide self-management education. In this study, all participants will participate in CHAMPION, but one arm will receive the experimental form (delivery via telehealth) and the other arm will receive the active comparator (delivery via telehealth).

SUMMARY:
The goal of this study is to evaluate the effectiveness of CHAMPION ("Comparative-effectiveness of a Healthy lifestyle and Asthma Management Program, In-person vs ONline"), a primary care-based intervention to address childhood obesity and asthma, and test the effectiveness of a telehealth-only version of the program. Intensive Health Behavior and Lifestyle Treatment (IHBLT), when delivered via telehealth vs. in-person among children with overweight or obesity and persistent asthma.

DETAILED DESCRIPTION:
This study will evaluate the comparative effectiveness of 1) telehealth delivery of CHAMPION vs. 2) in-person (standard of care) delivery of CHAMPION in a two-arm, individually randomized non-inferiority trial among 500 children. Obesity and asthma are two leading chronic diseases in children, and CHAMPION is an integration of the Healthy Weight Clinic (HWC) and pediatric Asthma Population Health Management Programming at Mass General Brigham. This study will address how to improve access to effective treatments consistent with United States Preventive Services Task Force (USPSTF) and American Academy of Pediatrics (AAP) guidelines that manage asthma and obesity concurrently in primary care among lower income diverse populations

ELIGIBILITY:
Caregiver-proxies will be 18 years old or older, English or Spanish speaking, and a primary caregiver of a child meeting the following criteria:

Inclusion criteria

* Age 4-17.9 years at time of screening
* BMI ≥ 85th percentile
* Asthma or reactive airway disease diagnosis, per child's Electronic Health Record (EHR) documentation and caregiver report

Exclusion criteria

* Diagnosis of anorexia nervosa, per child's EHR or caregiver report
* Pregnant, per child's EHR
* Plan to change pediatricians in the next year, per caregiver report
* Opted out of research, per child's EHR
* Sibling currently enrolled in the research trial, per enrollment log or caregiver report

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Child Body Mass Index (BMI) | 0-12 months
  Measured as BMI based on child height and weight
Change in Child BMI z-score | 0-12 months
  Measured as BMI based on child height and weight, and derived from Centers for Disease Control and Prevention (CDC) growth curves accounting for child age and sex
Change in Asthma Control Test | 0-12 months
  Per Asthma Control Test
Change in Asthma and Obesity Specific Quality of Life | 0-12 months
  Per response to caregiver-proxy survey

SECONDARY OUTCOMES:
Change in Child Diet Quality | 0-12 months
  Diet quality per Primescreen, via caregiver-proxy survey
Change in Child Average Hours of Sleep | 0-12 months
  Hours of sleep, via caregiver-proxy survey
Change in Child Average Days of Physical Activity | 0-12 months
  Days physically active for at least 60 minutes per day, via caregiver-proxy survey
Change in Child Average Hours of Screen Time | 0-12 months
  Hours of sedentary screen time, via caregiver-proxy survey
Asthma-related healthcare utilization | 0-12 months
  Per response to caregiver-proxy survey
Change in perceived stress (caregiver) | 0-12 months
  Per response to caregiver-proxy survey
Family-centered care assessment | 12 months
  Per response to caregiver-proxy survey
Telehealth satisfaction | 12 months
  Per response to caregiver-proxy survey
Barriers to program attendance | 12 months
  Per response to caregiver-proxy survey
Change in disordered eating symptoms | 0-12 months
  Per response to caregiver-proxy survey

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The funder, PCORI, requires data to be deposited into the Patient Centered Outcomes Data Repository/University of Michigan Inter-university Consortium for Political and Social Research (ICPSR).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be deposited after study completion.